CLINICAL TRIAL: NCT05867264
Title: Effect of Early Postoperative Oral Carbohydrate on Postoperative Recovery of the Unilateral Knee Arthroplasty: a Randomized, Single-blind, Parallel-controlled, Multicenter Study
Brief Title: Effect of Early Postoperative Oral Carbohydrate on Postoperative Recovery of the Unilateral Knee Arthroplasty
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hongwei Shi (Other)
Responsible Party: Sponsor-Investigator, Hongwei Shi, Director, Department of Anesthesiology, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nanjing First Hospital
Record Dates: First submitted 2023-04-08; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Oral Carbohydrates; Postoperative Recovery; Unilateral Knee Arthroplasty

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EOF 1 group：Early drinking water group (Placebo Comparator): After passing the evaluation by the anesthesiologist team in PACU, the EOF1 group drank 200ml of water.
  Interventions: Other: Early drinking water
- EOF 2 group: Early oral carbohydrate group (Experimental): After passing the evaluation by the anesthesiologist team in PACU, the EOF2 group had a drinking capacity of 200ml of 12.5% carbohydrates (100ml containing 12.5g of maltodextrin, fructose, and glucose).
  Interventions: Combination Product: Early consumption of carbohydrates
- Control group: Late feeding group (Placebo Comparator): After observing the vital signs for 30 minutes after surgery, patients in Group C were sent back to the ward to continue fasting and drinking for at least 6 hours. After the anus exhausts, they began to gradually drink and eat
  Interventions: Other: Late feeding group

INTERVENTIONS:
Other: Early drinking water — After passing the evaluation by the anesthesiologist team in PACU, the EOF1 group drank 200ml of water.
  The evaluation criteria for the anesthesiologist team are:
  1. Steward's awakening score is ≥ 6 points.
  2. Level of sobriety ≥ 3.
  3. There is no need to wait for intestinal peristalsis, based on the patient's wishes, and the feeding should be completed within 2 hours after the surgery.
  Arms: EOF 1 group：Early drinking water group
Combination Product: Early consumption of carbohydrates — After passing the evaluation by the anesthesiologist team in PACU, the EOF2 group had a drinking capacity of 200ml of 12.5% carbohydrates (100ml containing 12.5g of maltodextrin, fructose, and glucose).
  The evaluation criteria for the anesthesiologist team are:
  1. Steward's awakening score is 6 points.
  2. Level of sobriety ≥ 3.
  3. There is no need to wait for intestinal peristalsis, based on the patient's wishes, and the feeding should be completed within 2 hours after the surgery.
  Arms: EOF 2 group: Early oral carbohydrate group
Other: Late feeding group — After observing the vital signs for 30 minutes after surgery, patients in Group C were sent back to the ward to continue fasting and drinking for at least 6 hours. After the anus exhausts, they began to gradually drink and eat
  Arms: Control group: Late feeding group

SUMMARY:
To evaluate the effect of early postoperative oral carbohydrate on postoperative recovery of the unilateral knee arthroplasty

DETAILED DESCRIPTION:
Currently, most clinical studies on the impact of oral carbohydrates on postoperative recovery are focused on the preoperative stage, with only a few small sample studies indicating that postoperative oral carbohydrates can improve patient comfort. Orthopedic surgery, especially joint surgery, requires patients to start functional exercise as soon as possible after surgery. Joint replacement surgery requires reducing the consumption of muscle tissue caused by protein breakdown. Perioperative nutritional support for patients is of great significance for postoperative muscle function recovery and good functional exercise. However, further systematic research on the impact of early postoperative oral carbohydrates on postoperative recovery is still lacking.

This study selected patients who underwent unilateral total knee arthroplasty or single condylar arthroplasty. All surgical patients undergo homogenized preoperative preparation and intraoperative anesthesia management. Eligible patients were screened before surgery, and an informed consent form was signed. Patients enrolled in the experiment were randomly assigned into one of the three groups. They are the early feeding group (EOF1, EOF2group) and the late feeding group （control group）. Evaluate the effectiveness and safety of early postoperative feeding （EOF） in orthopedic surgery patients by measuring indicators such as insulin resistance index, QoR-15, and prealbumin and retinol binding protein.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79 years.
* Patients undergoing unilateral total knee arthroplasty or unicondylar joint replacement.
* Normal diet.
* ASA grade I~Ⅲ;
* BMI 18-30kg /m2.
* No intraspinal anesthesia contraindications.

Exclusion Criteria:

* Preoperative existence of gastric emptying disorders, such as gastrointestinal obstruction, gastroesophageal reflux, or previous gastrointestinal surgery.
* Patients with diabetes mellitus, severe renal dysfunction, or other severe metabolic diseases.
* History of motion sickness.
* Mental disorder, alcoholism, or a history of substance abuse.
* Patients with abnormal swallowing function.
* The operation time is greater than 3 hours.
* Maltodextrin fructose allergy or intolerance.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2023-05-25 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance index at fasting | 1 day after surgery
  In the venous blood in an early morning fasting state, the change in the insulin resistance index can reflect whether the carbohydrate administration is favorable in the early postoperative period.

SECONDARY OUTCOMES:
Insulin resistance index at fasting | on the day of the surgery
  In the venous blood in an early morning fasting state, the change in the insulin resistance index can reflect whether the carbohydrate administration is favorable in the early postoperative period.
Insulin resistance index at fasting | 3 days after surgery
  In the venous blood in an early morning fasting state, the change in the insulin resistance index can reflect whether the carbohydrate administration is favorable in the early postoperative period.
Pre albumin levels and retinol binding protein levels | on the day of surgery, 1 day and 3 days after surgery.
  The change in prealbumin levels and retinol-binding protein levels in venous blood in a fasting state in the early morning can reflect whether carbohydrate administration is favorable in the early postoperative period. Three of the eight test centers examined the pre-albumin levels and retinol-binding protein levels.
The 15-item recovery quality rating scale （QoR-15） | Up to 48 hours postoperative
  QoR-15 was used to assess five aspects of postoperative recovery quality (physical comfort, physical independence, psychological support, emotion and pain), with higher scores indicating the higher postoperative recovery quality. The lowest score is 0 points, and the highest score is 150 points.
The NRS score for the thirst thirst and hunger. | 2 hours, 6 hours and 8 hours after surgery
  The Numerical Rating Scale (NRS) is used to assess the degree of thirst and hunger in patients, with a score of 0 to 10. A score of 0 represents no thirst and no hunger, while a score of 10 represents unbearable thirst and hunger. The thirst and hunger score indicates that early postoperative carbohydrate administration is beneficial.
The degree of abdominal distension | 24 hours after surgery
  Using grading method, complaining of abdominal distention, tolerable, feeling gas rolling in the abdomen, no obvious abdominal signs, mild abdominal distension, abdominal distention, moderate abdominal distension, vomiting, dyspnea, and significant abdominal bulge.
Incidence of reflux aspiration and hypoxemia | 24 hours after surgery
  Reflux aspiration is defined as severe cough followed by hypoxemia and lung rale after vomiting. Hypoxemia is defined as SpO2<91% under air inhalation.
Anal exhaust time | Up to 48 hours postoperative
  The advanced time of the first postoperative anal exhaust indicates a favorable early postoperative carbohydrate administration.
Incidence of postoperative nausea and vomiting | Up to 48 hours postoperative
  The lower the incidence and severity of postoperative nausea and vomiting, indicating that early administration of carbohydrates after surgery is beneficial.
Hospitalization time | Up to 7days postoperative
  The shortened length of hospital stay indicated that early postoperative carbohydrate administration was advantageous.
The extent of the postoperative pain | Up to 48 hours postoperative
  The total amount of sufentanil consumed by the patient 48 hours after operation, the number of effective presses of the analgesia pump, the number of times of rescue analgesia and the amount of rescue drugs were converted into the total amount of morphine.
Patient satisfaction score | Up to 48 hours postoperative
  Rated on a 0-10 scale, with a higher score representing greater satisfaction.
The incidence and severity of various adverse events （AE） from the start of oral carbohydrates until the end of the trial | Up to 48 hours postoperative
  The lower the incidence and severity of various adverse events (AE) from the start of postoperative oral carbohydrates until the end of the trial, it indicates that the early postoperative carbohydrate administration is beneficial.
Number of antiemetic uses | Up to 24 hours after the first start of drug administration.
  The less use of antiemetic drugs within 24h after the first start of postoperative administration indicates that early postoperative carbohydrate administration is advantageous.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller TE, Roche AM, Mythen M. Fluid management and goal-directed therapy as an adjunct to Enhanced Recovery After Surgery (ERAS). Can J Anaesth. 2015 Feb;62(2):158-68. doi: 10.1007/s12630-014-0266-y. Epub 2014 Nov 13. PMID 25391735
- [Background] Rizvanovic N, Nesek Adam V, Causevic S, Dervisevic S, Delibegovic S. A randomised controlled study of preoperative oral carbohydrate loading versus fasting in patients undergoing colorectal surgery. Int J Colorectal Dis. 2019 Sep;34(9):1551-1561. doi: 10.1007/s00384-019-03349-4. Epub 2019 Jul 15. PMID 31309323
- [Background] Nygren J, Thorell A, Ljungqvist O. Preoperative oral carbohydrate therapy. Curr Opin Anaesthesiol. 2015 Jun;28(3):364-9. doi: 10.1097/ACO.0000000000000192. PMID 25827282
- [Background] Surgery Branch of Chinese Medical Association, Anesthesiology Branch of Chinese Medical Society. Chinese Expert Consensus and Path Management Guidelines for Accelerating Rehabilitation Surgery (2018) [J]. Chinese Journal of Anesthesiology, 2018,38 (001): 8-13.
- [Background] Yang R, Tao W, Chen YY, Zhang BH, Tang JM, Zhong S, Chen XX. Enhanced recovery after surgery programs versus traditional perioperative care in laparoscopic hepatectomy: A meta-analysis. Int J Surg. 2016 Dec;36(Pt A):274-282. doi: 10.1016/j.ijsu.2016.11.017. Epub 2016 Nov 10. PMID 27840308
- [Background] Bethune Orthopaedic Accelerated Rehabilitation Alliance, Bethune Charity Foundation Orthopaedic Professional Committee of trauma, Joint Surgery Professional Committee of Bethune Charity Foundation, etc. Guidelines for the management of perioperative fasting fasting in orthopaedic surgery [J]. Chinese Journal of Trauma and Orthopedics, 2019,21 (10): 829-834.
- [Background] Smith MD, McCall J, Plank L, Herbison GP, Soop M, Nygren J. Preoperative carbohydrate treatment for enhancing recovery after elective surgery. Cochrane Database Syst Rev. 2014 Aug 14;2014(8):CD009161. doi: 10.1002/14651858.CD009161.pub2. PMID 25121931
- [Background] Noba L, Wakefield A. Are carbohydrate drinks more effective than preoperative fasting: A systematic review of randomised controlled trials. J Clin Nurs. 2019 Sep;28(17-18):3096-3116. doi: 10.1111/jocn.14919. Epub 2019 Jun 10. PMID 31112338
- [Background] [9] Wang Cuilan, Huang Yuting, Zeng Qing, et al. Study on postoperative fasting water prohibition time under ERAS concept [J]. Clinical Medical Engineering, 2022,29 (4): 2.

DOCUMENTS (1):
  • Study Protocol (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT05867264/Prot_000.pdf